CLINICAL TRIAL: NCT04437810
Title: To Study Efficacy of Albumin in Cirrhosis With Spontaneous Bacterial Peritonitis at Low Risk for AKI Development - A Randomised Placebo Controlled Trial- A Pilot Study
Brief Title: To Study Efficacy of Albumin in Cirrhosis With Spontaneous Bacterial Peritonitis at Low Risk for AKI Development
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-31
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Liver Cirrhosis; Acute Kidney Injury
MeSH Terms: conditions — Liver Cirrhosis; Acute Kidney Injury | interventions — Albumins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin+ SMT (Experimental): Patients in the Albumin Arm will receive Human Albumin 20% 1.5g/kg body weight (Maximum 100g) within 6 hours from the time of diagnosis over a period of 12 hours, followed by 1g/kg bodyweight (Maximum 100g) over a period of 12 hours after 48 hours of diagnosis.(D3) along with standard medical therapy
  Interventions: Biological: Albumin; Other: Standard Medical Treatment
- Placebo+SMT (Placebo Comparator): - Patients in placebo arm will receive similar volume of isotonic fluid (saline) over same duration of time along with standard medical therapy
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Biological: Albumin — - Patients in the Albumin Arm will receive Human Albumin 20% 1.5g/kg body weight (Maximum 100g) within 6 hours from the time of diagnosis over a period of 12 hours, followed by 1g/kg bodyweight (Maximum 100g) over a period of 12 hours after 48 hours of diagnosis.(D3)
  Arms: Albumin+ SMT
Other: Standard Medical Treatment — standard medical therapy

SUMMARY:
The role of Albumin in prevention and Treatment of Acute Kidney Injury (AKI) in patients with Spontaneous Bacterial Peritonitis (SBP) who are at high risk of AKI development has been clearly defined , which decreases the morbidity and mortality. But the role of Albumin in patient with SBP who are at low risk of AKI development (Serum Bilirubin <4mg/dl, Creatinine <1mg/dl at the time of presentation) has been controversial and there are no placebo controlled trials. We propose that Albumin at the standard doses is beneficial in preventing development of AKI in patients with SBP who are at low risk of AKI development.

DETAILED DESCRIPTION:
1. Aim- To compare the efficacy of albumin when compared to placebo in the development or progression of AKI in patients with cirrhosis and spontaneous bacterial peritonitis who are at low risk for AKI development (i.e Serum Bilirubin <4 mg/dL and serum creatinine < 1 mg/dl at presentation)

   * Primary objective: To evaluate the Proportion of patients developing AKI by day 7
   * Secondary objectives:
   * To compare the resolution of SBP by day 2 and day 5 in both the groups
   * To measure the Changes in PRA, TNF-α, IL-6 at day 7
   * To measure the Changes in renal resistive index at day 7
   * To compare Mortality by day 7 and 28 in both the groups
2. Methodology:

   1. Dose and duration of albumin/placebo infusion in both the limbs: -The dose of albumin was 1.5 g/kg of body weight given within 6 h of SBP being diagnosed over a period of 12hrs, followed by an additional infusion of 1.0 g/kg on day 3 over a period of 12 hrs. Other arm receives a similar quantity of isotonic fluid like normal saline or plasmalyte
   2. Renal resistive index will be done with the help of a) high frequency probe(5Mhz) together with the use of color or power Doppler to help vessel localization., sampling for RRI should be done at the level of the arcuate or interlobar arteries, adjacent to medullary pyramids. Measurements will be repeated in different parts of both organs (superior, median, and lower) when at least three reproducible waveforms have been obtained. An RRI will be calculated with the following formula: (peak systolic velocity - end diastolic velocity)/peak systolic velocity, and the mean value of three measurements at each kidney will be considered. An RRI value 0.60 ± 0.01 (mean ± SD) is usually taken as normal with a value of 0.70 being considered the upper normal threshold by most authors. In order to maximize waveform size, care will be taken in using the lowest pulse repetition frequency without aliasing, the highest possible gain without noise and the lowest wall filter. Patient will undergo RRI on day 0 and day 7.
   3. PRA, TNF-A and IL-6: - Measurement at day 0 and day 7 PRA is measured by generating AngI (angiotensin I) from endogenous angiotensinogen, followed by measurement by RIA of the generated AngI. Although PRA measurement is convenient for estimating the biological activity of the renin system, it may not necessarily reflect the real concentration of active renin. Il-6 is measured with the help of IL-6 ELISA kits. TNF- alpha is measured using flow cytometry.
   4. Antibiotics to be used in the SBP: - The gold standard treatment consists of third-generation cephalosporins, especially cefotaxime/ceftriaxone, given intravenously at a dose of 4-8 g/d for a minimum duration of 5 d. (AASLD guidelines). If patient does not respond then switch over to carbapenem (meropenem) with or without tigecycline. if patient still does not respond then GM-CSF will be given.
   5. Blood samples and Ascitic fluid samples will be collected and stored for measurement of Neutrophilic activity (CD66+/CD66-, CD11b) and Macrophage activity (CD 14+, CD 16+, IL-6, TNF-α)
   6. Serum Cystatin C and Urinary NGAL, markers and predictors of renal injury will be measured in both the limbs.

      Management of the complications: -
      * The patients who develop sepsis (presence of SIRS; positive blood cultures); worsening of hepatic encephalopathy >2 grades, variceal bleed or deterioration of the clinical condition; worsening of AKI and volume overload will be managed according to standard protocols,
      * Definitions: -
      * Spontaneous bacterial peritonitis: - SBP was diagnosed when the ascitic fluid polymorphonuclear (PMN) cell count was > 250 cells/mm3.
      * Resolution of Spontaneous bacterial peritonitis: - A repeat diagnostic paracentesis to document the response by a greater-than 25% decrease in ascitic fluid neutrophil count at 48 h after initiation of antibiotics is recommended

      Study population: Patients with Cirrhosis of Liver who presents with Spontaneous Bacterial Peritonitis with baseline creatinine <1mg/dl and Serum Bilirubin <4mg/dl

      Study Design: Single Center, Double Blinded (Patient and Treating physician), Placebo Controlled (Saline), Randomised Controlled Trial- a pilot study

      Study period: 1.5 year from the date of ethics approval (2020-2022)

      Sample size with justification: The study will be conducted as a pilot study and all the cases with SBP with low risk for AKI development will be recruited. The minimum number of subjects expected to be enrolled is 100.

      Intervention:
      * Patients in the Albumin Arm will receive Human Albumin 20% 1.5g/kg body weight (Maximum 100g) within 6 hours from the time of diagnosis over a period of 12 hours, followed by 1g/kg bodyweight (Maximum 100g) over a period of 12 hours after 48 hours of diagnosis.(D3) along with Standard medical therapy
      * Patients in placebo arm will receive similar volume of isotonic fluid (saline) over same duration of time along with standard medical therapy
      * Monitoring and assessment:

      This RCT will be conducted at ILBS New Delhi

      The following data will be recorded for each patient:
      * Etiology of cirrhosis, duration, Large volume paracentesis
      * H/o of jaundice, distension abdomen, swelling feet, altered sensorium, vomiting of blood or passing melena
      * Height, weight and BMI
      * Investigations: CBC, LFT, PT/INR, KFT.
      * Disease severity (CTP and MELD scores)
      * Day 0 - Hemogram, prothrombin time/ INR, KFT, LFT, TNF alpha,IL-6, PRA, ABG, blood culture, urine culture, chest X-ray, urine R/M, ascitic fluid analysis for the TLC, DLC, sugar, protein, albumin, culture, gram stain and Urine NGAL and Serum cystatin C ,Renal Resistive Index(RRI) will be done and ECG, ECHO for the volume overload, IVC diameter.
      * DAY 2 - hemogram, KFT, LFT, ABG, chest X-ray, and ascitic fluid analysis for the TLC, DLC, culture, gram stain
      * DAY 7: - PRA, TNF-alpha, IL-6
      * DAY 7: - Renal Resistive Index,
      * Day 28-- hemogram, prothrombin time/ INR, KFT, LFT
      * Statistical Analysis:
      * Continuous variables- Mean +/- SD
      * Categorical variables as percentages (%) or Frequencies
      * Student t test will be applied in continuous data compared with two groups
      * Survival analysis like Cox-Regression model and Kaplan-Meir plots will be plotted to find the possible factors responsible for mortality
      * Besides these, Intent to treat (ITT) and Per Protocol (PP) will be done at the time of data analysis.

      Adverse effects:
      * Patients receiving Albumin may experience Nausea, Vomiting, Fever with chills, dyspnea Wheezing, Volume overload, Anaphylactic reaction
      * Stopping rule of study:
      * In Albumin arm

        * Development of AKI
        * Adverse reaction to drug
        * Cardiopulmonary compromise
      * In Placebo Arm

        * Development of AKI
        * Development of Septic Shock

ELIGIBILITY:
Inclusion Criteria:

* Patients who are above 18 years of age
* Patients with Cirrhosis and SBP (community acquired /Health care associated/ nosocomial) with baseline Creatinine <1mg/dl, Bilirubin <4mg/dl

Exclusion Criteria:

* Antibiotic treatment within one week before the diagnosis of SBP (except for prophylactic treatment with norfloxacin)
* Significant cardiac failure, pulmonary disease
* Known Chronic Kidney Disease or findings suggestive of organic nephropathy (proteinuria, haematuria, or abnormal findings on renal USG)
* Hepatocellular carcinoma
* HIV infection;
* GI bleed within 1 month before the study
* Ileus
* Grade 3 to 4 hepatic encephalopathy
* Other types of infection
* Shock
* Serum Bilirubin ≥4 mg/dL and Serum Creatinine ≥ 1 mg/dl at presentation
* Patients requiring Albumin for any other indication.
* Presence of any potential causes of dehydration (such as diarrhea or an intense response to diuretic treatment) within one week before the diagnosis of SBP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients having development / progression of Acute Kidney Injury in both groups. | Day 7

SECONDARY OUTCOMES:
Resolution of Spontaneous Bacterial Peritonitis in both groups | Day 2
  Ascitic fluid absolute neutrophil count < 250
Resolution of Spontaneous Bacterial Peritonitis in both groups | Day 7
  Ascitic fluid absolute neutrophil count < 250
Change in PRA in both groups | Day 7
Change in TNF-alpha in both groups | Day 7
Change in IL-6 in both groups | Day 7
Change in Renal resistive index in both groups | Day 7
Mortality in both groups | Day 7
Mortality in both groups | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided